CLINICAL TRIAL: NCT01841775
Title: Pharmacovigilance Study of the Interferon α 2b Produced by Bio-Manguinhos / Fiocruz and Used by Genotype 2/3 Chronic Hepatitis C Patients (Estudo de farmacovigilância da Alfainterferona 2b Humana Recombinante Produzida Por Bio-Manguinhos - Fiocruz, Utilizada em Portadores de Hepatite C crônica genótipos 2 e 3 Atendidos Pelo Programa de Medicamentos de Dispensação em Caráter Excepcional no Estado do Rio de Janeiro)
Brief Title: Interferon α 2b Pharmacovigilance Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Collaborators: Hospital Federal de Bonsucesso (Bonsucesso Federal Hospital) (Unknown); Hospital Universitário Clementino Fraga Filho (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIGAT-RJ IFNα2b
Record Dates: First submitted 2013-04-19; First posted 2013-04-29 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C, Chronic; Genotype 2/3; Interferon α 2b; Ribavirin; Pharmacovigilance
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: interferon α 2b + ribavirin — 1. interferon α 2b: 3.000.000 IU SUBQ 3 times / wk for 24 weeks
  2. ribavirin 250 mg: 15mg/kg/day,ORALLY twice a day for 24 weeks

SUMMARY:
Multicenter prospective follow-up of a not controlled chronic hepatitis C genotypes 2/3 patients cohort with treatment indication with interferon α 2b and ribavirin for 24 weeks, and the verification of sustained virological response at week 48.

The eligibility criteria and outcome measures followed the Clinical Protocol and Therapeutic Guidelines for Chronic Viral Hepatitis C, published by the Ministry of Health:

http://portal.saude.gov.br/portal/arquivos/pdf/pcdt_hepatite_c_2011_retificado.pdf

ELIGIBILITY:
Inclusion Criteria:

* Genotype 2/3 Chronic Hepatitis C confirmed by biomolecular technology (RNAVHC);
* Treatment naive;
* Signing the Informed Consent Form;
* Eligibility criteria and outcome measures followed the Clinical Protocol and Therapeutic Guidelines for Chronic Viral Hepatitis C, published by the Ministry of Health: http://portal.saude.gov.br/portal/arquivos/pdf/pcdt_hepatite_c_2011_retificado.pdf

Exclusion Criteria:

* Serious adverse events;
* Intolerance to treatment;
* Lost to follow up.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2009-05; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Adverse events | Up to 24 weeks
  * Diary for recording adverse events by patients daily;
  * Monthly follow-up interview with MD and PharmD

SECONDARY OUTCOMES:
Sustained virological response | 24 weeks after finishing treatment

CONTACTS AND LOCATIONS:
Overall Officials: Eliane M. dos Santos, MD, MSc, Principal Investigator — The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz); Paulo Roberto G. dos Santos, PharmD, MSc, Study Director — The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz); Deborah A. da Conceição, BScN, Study Director — The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz)
Locations (2):
- Brazil (2):
  - Hospital Federal de Bonsucesso (Bonsucesso Federal Hospital), Rio de Janeiro, Rio de Janeiro
  - Hospital Universitário Clementino Fraga Filho (Clementino Fraga Filho University Hospital), Rio de Janeiro, Rio de Janeiro